CLINICAL TRIAL: NCT00891995
Title: Effect of Metabolic Control at Onset of Diabetes on Progression of Type 1 Diabetes
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Primary outcome evaluation determined lack of treatment group difference
Sponsor: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DirecNet 012; NCT00505206 (obsolete NCT alias)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Closed Loop Therapy; Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Glucose Self-Monitoring; Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensive Treatment (Experimental): closed loop therapy (4-6 days), insulin pump (2 years), continuous glucose monitoring (2 years), home glucose monitoring (2 years)
  Interventions: Device: Closed loop; Device: Home glucose monitoring; Device: Insulin pump; Device: Continuous glucose monitor
- Standard Treatment (Active Comparator): home glucose monitoring (2 years)
  Interventions: Device: Home glucose monitoring

INTERVENTIONS:
Device: Closed loop — Closed loop therapy for up to 4 to 6 days
  Arms: Intensive Treatment
Device: Home glucose monitoring — Standard diabetes management using a home glucose meter.
Device: Insulin pump — Insulin pump use for 2 years
  Arms: Intensive Treatment
Device: Continuous glucose monitor — Continuous glucose monitor use for 2 years
  Arms: Intensive Treatment

SUMMARY:
The purpose of this study is to find out if very tight blood glucose control from the onset of Type 1 Diabetes can preserve beta cell function. Study subjects will be randomly assigned to receive either standard diabetes management or intensive diabetes management, which involves several days of closed loop therapy followed by home use of a continuous glucose monitor and insulin pump.

DETAILED DESCRIPTION:
The specific aim of this study is to determine if early restoration of metabolic control will improve C-peptide production compared to children receiving routine diabetes management and the secondary aim is to determine if allowing the islet cells to be less metabolically active will have an impact on the underlying autoimmune process.

Following completion of the baseline procedures (Mixed Meal Tolerance Test and blood sample collection), participants are randomized to either the Standard Treatment Group or the Intensive Treatment Group which includes 4-6 days of inpatient closed loop therapy followed by outpatient use of an insulin pump and continuous glucose monitor for diabetes management.

All subjects will be seen 7 times in the first year and 4 times in the second year for follow-up testing. Subjects who are still producing insulin after 2 years may be asked to return every 6 months for an additional 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 6.0 to <46.0 years
* Diagnosis of type 1 diabetes with initiation of insulin therapy within past 7 days (day 1 being the first day of insulin therapy)
* If participant is female with reproductive potential, willing to avoid pregnancy and pregnancy test negative.
* Willing to accept randomization to either the intensive diabetes management group or the standard care group.
* Willing to complete the planned 2 years of follow-up.
* Able to electronically transmit data monthly.
* Investigator believes that the participant (and parent/guardian for children) understands and agrees to comply with the study protocol and is capable of undertaking all necessary testing.

Exclusion Criteria:

* Currently pregnant or lactating, or anticipate getting pregnant in the next one year.
* Currently anemic (hematocrit level will be obtained at the screening visit).
* Chronic use of systemic steroids or other noninsulin pharmaceuticals that might affect glycemic control or the presence of a disease that is likely to be treated with such medications during the first two years of the study.
* Complicating medical issues that might interfere with study conduct.
* Inpatient psychiatric treatment in the past 6 months (if the participant is a minor, for either the participant or the participant's primary care giver).
* Currently participating in another type 1 diabetes treatment study, including an intervention trial for treatment of diabetic ketoacidosis.

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy W Beck, M.D., Ph.D., Study Director — Jaeb Center for Health Research; Jay S. Skyler, M.D., M.A.C.P., Principal Investigator — University of Miami
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Indiana University, Indianapolis, Indiana
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Background] Buckingham B, Beck RW, Ruedy KJ, Cheng P, Kollman C, Weinzimer SA, DiMeglio LA, Bremer AA, Slover R, Tamborlane WV; Diabetes Research in Children Network (DirecNet) Study Group; Type 1 Diabetes TrialNet Study Group. Effectiveness of early intensive therapy on beta-cell preservation in type 1 diabetes. Diabetes Care. 2013 Dec;36(12):4030-5. doi: 10.2337/dc13-1074. Epub 2013 Oct 15. PMID 24130350
- [Result] Diabetes Research in Children Network (DirecNet) Study Group; Type 1 Diabetes TrialNet Study Group; Buckingham BA, Beck RW, Ruedy KJ, Cheng P, Kollman C, Weinzimer SA, DiMeglio LA, Bremer AA, Slover R, Cantwell M. The effects of inpatient hybrid closed-loop therapy initiated within 1 week of type 1 diabetes diagnosis. Diabetes Technol Ther. 2013 May;15(5):401-8. doi: 10.1089/dia.2013.0002. Epub 2013 Apr 9. PMID 23570538

RESULTS

PARTICIPANT FLOW:
Groups:
- Intensive Treatment: The Intensive Treatment group will participate in 4-6 days of inpatient closed loop therapy followed by use of an insulin pump and continuous glucose monitoring (CGM) in addition to standard monitoring with a home glucose meter for 2 years.
- Standard Treatment: The Standard Care group will receive standard diabetes management using a home glucose meter for blood sugar monitoring for 2 years.
Period: Overall Study
Arm/Group | Intensive Treatment | Standard Treatment
Started | 50 | 21
Completed | 50 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only 48 participants in the intensive treatment group and 20 participants in the standard treatment group who show any positive autoantibody in the first year were included in the analyses.
Groups:
- Intensive Treatment: The Intensive Treatment group will participate in 4-6 days of inpatient closed loop therapy followed by use of an insulin pump and CGM in addition to standard monitoring with a home glucose meter for 2 years.
- Total: Total of all reporting groups
Arm/Group | Intensive Treatment | Standard Treatment | Total
Number analyzed (Participants) | 48 | 20 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 19 | 65
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (4.7) | 14.7 (7.6) | 13.3 (5.7)
Gender [Count of Participants; unit: Participants]
  Female | 17 | 7 | 24
  Male | 31 | 13 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  White | 42 | 18 | 60
  Black | 1 | 0 | 1
  Hispanic or Latino | 2 | 1 | 3
  More than one race | 1 | 0 | 1
  Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: C-peptide Average Area Under the Curve (AUC) in Response to a Mixed Meal at 1 Year Following Enrollment.
Description: In the primary analysis of the 12-month Mixed-Meal Tolerance Test (MMTT) results, the geometric mean (95% C.I.) of C-peptide average AUC (=AUC/time) was 0.43 (0.34, 0.52) pmol/ml in the intensive treatment group and 0.52 (0.32, 0.75) pmol/ml in the usual care group (P=0.49).
Time Frame: At baseline, MMTT data were collected at 0 and 90 min; at 12 months, MMTT data were collected at 0 to 240 min post meal
Population: Among the 68 participants who completed 1 year visit and with positive autoantibody, 1 participant in the intensive treatment group did not complete MMTT test, thus was excluded from all C-peptide analyses.
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/ml
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 47 | 20
pmol/ml | 0.43 [0.34 to 0.52] | 0.52 [0.32 to 0.75]
Statistical Analysis 1: Comparison: Intensive Treatment vs Standard Treatment; Test type: Superiority or Other; p = 0.49, ANCOVA — One-sided p-value; Adjusted for baseline C-peptide AUC, age, gender and diabetic ketoacidosis

2. Secondary Outcome: Peak C-peptide in Response to a Mixed Meal at 1 Year Following Enrollment
Time Frame: 0 to 240 min post meal at 1 year MMTT
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/ml
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 47 | 20
pmol/ml | 0.53 [0.42 to 0.65] | 0.65 [0.40 to 0.95]

3. Secondary Outcome: Incidence of the Loss of the 2 Hour Peak C-peptide < 0.2 Pmol/ml on a Semi-annual MMTT
Description: Outcome measure in the table is the incidence of 2 hour peak C-peptide>=0.2 pmol/ml. Since the formal clinical trial stopped at 12 months due to lack of efficiency (later follow-up were used to collect data for secondary analyses by pooling the two groups), only the outcome at 12 months are reported.
Time Frame: 0 to 240 min post meal at 1 year MMTT
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 47 | 20
participants | 37 | 16

4. Secondary Outcome: HbA1c
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 48 | 20
percent | 7.4 (1.2) | 7.3 (1.1)
Statistical Analysis 1: Comparison: Intensive Treatment vs Standard Treatment; Test type: Superiority or Other; p = 0.40, ANCOVA — One-sided p-value; Adjusted for baseline A1c, age, gender and Diabetic ketoacidosis

5. Secondary Outcome: Adverse Events (Severe Hypoglycemia)
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 48 | 20
participants | 1 | 0

6. Secondary Outcome: CGM Mean Glucose
Time Frame: 1 year
Population: Participants who used CGM (either blinded or unblinded CGM) for at least 24 hours at 12 months.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 31 | 15
mg/dL | 150 [117 to 186] | 152 [145 to 171]

7. Secondary Outcome: CGM Measured Glucose Outcomes
Description: Include a series of glucose indices created from CGM measured glucose data, such as % time with glucose values <=70 mg/dl, % time with glucose values within target range of 71-180 mg/dl, % time with glucose values >180 mg/dl, and glucose variability as measured by coefficient of variation. These indices were calculated by giving equal weight to each of the 24 h of the day. At least 24 h of CGM data were required for calculating these indices.
Time Frame: 1 year
Population: Participants who used CGM (either blinded or unblinded CGM) for at least 24 hours at 12 months.
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 31 | 15
percent
  %Glucose 71-180 mg/dL | 69 [47 to 83] | 70 [57 to 79]
  %Glucose <=70 mg/dL | 2.5 [0.4 to 7.7] | 0.7 [0.0 to 5.0]
  %Glucose >180 mg/dL | 27 [8 to 49] | 22 [18 to 41]
  %Coefficient of variation | 35 [29 to 39] | 35 [28 to 38]

8. Secondary Outcome: Daily Insulin Dose
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: u/day/kg
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 48 | 20
u/day/kg | 0.6 (0.2) | 0.6 (0.3)

9. Secondary Outcome: BMI Percentile
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Intensive Treatment | Standard Treatment
Number analyzed (Participants) | 46 | 19
percent | 58 [39 to 81] | 62 [40 to 72]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intensive Treatment | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 2/48 | 1/20
Other Adverse Events (participants affected / at risk) | 6/48 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Treatment (N=48) | Standard Treatment (N=20)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — In the usual care group, one participant was hospitalized for gastroenteritis.
Anaphylactic reaction (General disorders) | 1 (1) | 0 (0) — During inpatient hybrid closed-loop control (HCLC) therapy, one subject had an anaphylactic reaction following his first dinner, presumably resulting from a peanut allergy, and received intravenous steroids.
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) — During follow up, in the intensive group, one participant with a prior history of depression developed suicidal ideation.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensive Treatment (N=48) | Standard Treatment (N=20)
severe hypoglycemia (Endocrine disorders) | 1 (2) | 0 (0) — Severe hypoglycemia occurred in one participant (two events, at 6 months while CGM was being used and 12 months after CGM had been discontinued) in the intensive group and in no participants in the usual care group.
venous thrombosis (Vascular disorders) | 2 (2) | 0 (0) — There were two cases of venous thrombosis related to the intravenous line that resolved without consequence.
faint (General disorders) | 1 (1) | 0 (0) — During follow up, in the intensive group, one participant fainted following the 3-month MMTT
skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — During follow up, in the intensive group, one participant had a skin infection related to the CGM sensor insertion.
depression and anxiety (Psychiatric disorders) | 0 (0) | 2 (2) — In the usual care group, two participants developed depression and anxiety.
Needle stick/puncture (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — On admission, during insertion of sensor into abdomen of patient, the skin was pinched up due to minimal body fat. The sensor entered subject's skin then exited other side and punctured nurse's thumb which resulted in cross contamination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No